CLINICAL TRIAL: NCT00968227
Title: Effect of Red Blood Cell Transfusion on Brain Metabolism in Patients With Subarachnoid Hemorrhage
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-0733; NIH 5P50NS035966-10
Record Dates: First submitted 2009-08-26; First posted 2009-08-28 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Subarachnoid Hemorrhage; Vasospasm
Keywords: subarachnoid hemorrhage; vasospasm; transfusion; cerebral oxygen delivery; hemoglobin
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Erythrocyte Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transfusion (Experimental)
  Interventions: Biological: Red blood cell transfusion

INTERVENTIONS:
Biological: Red blood cell transfusion — Transfusion of 1 unit of packed red blood cells over 1 hour.

SUMMARY:
The purpose of this study is to determine if giving blood transfusions to anemic patients with subarachnoid hemorrhage will reduce their chances of having a stroke from vasospasm.

DETAILED DESCRIPTION:
Each year, approximately 30,000 people suffer aneurysmal subarachnoid hemorrhage (SAH) in the United States. The most common and potentially treatable cause of secondary neurological injury in this population is delayed ischemic deficit (DID). As the name implies, this phenomenon is fundamentally a reduction of cerebral blood flow (CBF) and oxygen delivery below critical ischemic thresholds, occurring days after the onset of hemorrhage. Three inter-related physiological processes appear to be involved in the reduced oxygen delivery: severe narrowing of intracranial arteries (arterial vasospasm), intravascular volume depletion and a loss of normal autoregulatory function in the distal circulation. DID occurs in up to 40% of patients surviving SAH. One third of these patients will die from this phenomenon and another third will be left with permanent and severe disability.

The optimal treatment of vasospasm is not known. Medical management involves a number of hemodynamic manipulations and is usually referred to as hypervolemic, hypertensive, hemodilution (or Triple-H) therapy. Our knowledge of the physiological impact of the individual components or a combination of them is limited and clinical efficacy has not been established. The information gained in this study has great potential to advance our knowledge regarding the role of hematocrit in the optimal treatment of this often-devastating condition.

Changes in hematocrit can potentially impact brain oxygen delivery in two ways. First, there is a linear relationship between hemoglobin and arterial oxygen content, lower hematocrit less oxygen. Thus at a given CBF lowering hematocrit reduces brain oxygen delivery. Fortunately, the brain responds to this by increasing blood flow to restore oxygen delivery to baseline levels. Additionally, lowering hematocrit has another effect, it reduces viscosity which in and of itself can raise CBF, but in a non-linear way. It is the relative contribution of these two effects that will determine if oxygen delivery improves.

It has been proposed by largely on theoretical consideration that the "optimal" hematocrit that achieves this balance is 30-35%. Yet no study to date has assessed the relationship between hematocrit and oxygen delivery in SAH patients. Other observations, however, suggest that higher hemoglobin levels in SAH patients was associated with better outcomes. Finally another retrospective review suggested that receiving transfusions increased risk for vasospasm and poor outcome after subarachnoid hemorrhage.

We are proposing to begin a series of studies to determine the appropriate management of hematocrit in SAH patients. The first is to define the appropriate physiologic response (cerebral oxygen delivery and metabolism) to a change in hematocrit. Then the "optimal" hematocrit can be defined. Only then will we be able to properly design clinical outcome trials.

ELIGIBILITY:
Inclusion Criteria:

1. Aneurysmal SAH confirmed by angiography
2. Hemoglobin < 12.5 gm/dl
3. One of the following:

   * Considered at increased risk for vasospasm by care team
   * Angiographic vasospasm
   * Delayed ischemic deficit
4. Able to be studied within 2 weeks after subarachnoid hemorrhage

Exclusion Criteria:

1. Active Coronary Artery Disease
2. Severe congestive heart failure
3. Jehovah's witness
4. Unable to obtain appropriately matched blood
5. Other contraindications for transfusion
6. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-11; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Diringer, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University Medical Center, St Louis, Missouri, United States

REFERENCES:
- [Result] Dhar R, Zazulia AR, Videen TO, Zipfel GJ, Derdeyn CP, Diringer MN. Red blood cell transfusion increases cerebral oxygen delivery in anemic patients with subarachnoid hemorrhage. Stroke. 2009 Sep;40(9):3039-44. doi: 10.1161/STROKEAHA.109.556159. Epub 2009 Jul 23. PMID 19628806

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transfusion
Started | 56
Completed | 56
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Transfusion
Number analyzed (Participants) | 56
Age, Continuous [Mean (Full Range); unit: years] | 54 [48 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 44
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 56

OUTCOME MEASURES:

1. Primary Outcome: Change in Oxygen Delivery in Vulnerable Brain Regions
Description: Change in oxygen delivery after transfusion in brain regions with low baseline delivery.
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: ml/100g/min
Arm/Group | Transfusion
Number analyzed (Participants) | 47
ml/100g/min
  Baseline | 3.7 (0.5)
  Post transfusion | 4.3 (0.9)
Statistical Analysis 1: Comparison: Transfusion; Test type: Superiority — Paired t-test; p = 0.001, t-test, 2 sided

2. Secondary Outcome: Change in Oxygen Extraction Fraction in Regions With Low Baseline Delivery.
Description: Change in oxygen extraction fraction after transfusion of 1 unit of RBC in regions with low baseline delivery (DO2 < 4.5 ml/100g/min.
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: fraction
Arm/Group | Transfusion
Number analyzed (Participants) | 34
fraction
  Baseline | 0.49 (0.14)
  Post transfusion | 0.44 (0.14)

ADVERSE EVENTS:
Arm/Group | Transfusion
All-Cause Mortality (participants affected / at risk) | 4/56
Serious Adverse Events (participants affected / at risk) | 0/56
Other Adverse Events (participants affected / at risk) | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No